CLINICAL TRIAL: NCT05297214
Title: A Study of Acute Kidney Injury in Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Abdelsabour Hassan, resident doctor at pediateric department sohag General hospital, Sohag University
Other Study IDs: soh-Med-22-03-11
Record Dates: First submitted 2022-03-13; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Cell Count; Kidney Function Tests; Blood Gas Analysis; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum creatinine and Other investigations will be done according to the case — following up AKI patients with serum creatinine,Urine out put, CBC,Serum electrolytes,renal functin test,Liver function test,urine analysisand specific investigations according to case
  Other Names: complete blood count, kidney function tests, blood gases, serum electrolytes, and urine analysis,abdominal ultrasound, others according to case as C3,c4,ANA,ANCA,AntidsDNA,Protein creatinin ratio

SUMMARY:
Acute kidney injury (AKI) has been traditionally defined as an abrupt loss of kidney function leading to a rapid decline in the glomerular filtration rate (GFR), accumulation of waste products such as blood urea nitrogen (BUN) and creatinine, and dysregulation of extracellular volume and electrolyte homeostasis . Acute kidney injury (AKI) is a very common condition, especially among hospitalized patients.

this work aims to study the demographics, etiology, clinical characteristics, and outcome of acute kidney injury in children in Sohag University Hospital - Pediatrics Department.

ELIGIBILITY:
Inclusion Criteria:

* All children with acute kidney injury with an age range from 1 month to 16 years old

Exclusion Criteria:

1. patients with chronic kidney disease (CKD)
2. Patients with irregular follow up
3. Patients with incomplete data
4. Patients whose medical guardians refuse participation in the study

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: Acute kidney injury (AKI) will be defined by the presence of an Increase in serum creatinine by 0.3 mg/dL or more within 48 hours, or increase in serum creatinine to 1.5 times or more baseline within the prior seven days, or urine output less than 0.5 mL/kg/h for at least 6 hours . AKI will be classified according to serum creatinine level (SCr) and urine output as in table .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine level | one year
  follow up AKI patients with serum creatinine level

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag General Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tresa V, Yaseen A, Lanewala AA, Hashmi S, Khatri S, Ali I, Mubarak M. Etiology, clinical profile and short-term outcome of acute kidney injury in children at a tertiary care pediatric nephrology center in Pakistan. Ren Fail. 2017 Nov;39(1):26-31. doi: 10.1080/0886022X.2016.1244074. Epub 2016 Oct 21. PMID 27767356
- [Background] Akcay A, Turkmen K, Lee D, Edelstein CL. Update on the diagnosis and management of acute kidney injury. Int J Nephrol Renovasc Dis. 2010;3:129-40. doi: 10.2147/IJNRD.S8641. Epub 2010 Sep 29. PMID 21694939
- [Background] Lameire NH, De Vriese AS, Vanholder R. Prevention and nondialytic treatment of acute renal failure. Curr Opin Crit Care. 2003 Dec;9(6):481-90. doi: 10.1097/00075198-200312000-00004. PMID 14639067
- [Background] Kaddourah A, Basu RK, Bagshaw SM, Goldstein SL; AWARE Investigators. Epidemiology of Acute Kidney Injury in Critically Ill Children and Young Adults. N Engl J Med. 2017 Jan 5;376(1):11-20. doi: 10.1056/NEJMoa1611391. Epub 2016 Nov 18. PMID 27959707